CLINICAL TRIAL: NCT05440110
Title: Cognitive Effects and Potential Mechanisms of Theta-burst Stimulation (TBS) in Suspected Non-Alzheimer Disease Pathophysiology (SNAP): a Pilot Study
Brief Title: Cognitive Effects of Theta-burst Stimulation (TBS) in Suspected Non-Alzheimer Disease Pathophysiology (SNAP)
Acronym: SNAP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202200400A0
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Suspected Non-Alzheimer Disease Pathophysiology (SNAP)
Keywords: Suspected Non-Alzheimer Disease Pathophysiology (SNAP); theta-burst stimulation; repetitive transcranial magnetic stimulation (rTMS)

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized controlled clinical trial for the first two weeks, followed by an open-label trial for the next two weeks, and combined functional neuroimaging study of 18F-FDG-PET to further explore the potential mechanisms. A total of 20 SNAP dementia patients will be recruited for consecutive two years, and be subjected to iTBS for 5 daily interventions per week for four consecutive weeks. Cognitive evaluation will be performed before and immediately after TBS intervention, and 8 weeks after TBS. Data on functional neuroimaging will be also collected before and after TBS protocol.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active and active (Active Comparator): The patients will be subjected to TBS for 5 daily interventions per week for four consecutive weeks.
  Interventions: Device: active and active TBS
- sham and active (Sham Comparator): The patients will be subjected to TBS for 5 daily interventions per week for the first two weeks, followed by an open-label trial for the next two weeks.
  Interventions: Device: sham and active TBS

INTERVENTIONS:
Device: active and active TBS — The investigators will perform standard intermittent TBS (iTBS) parameters to left DLPFC of every patient in the study. The frequency parameters of TBS are 3-pulse 50- Hz bursts, every 200 ms at 5 Hz, and the intensity is 90% of active motor threshold. A single session of iTBS contains 2 s of TBS repeated every 10 s for 20 times. In this study, The investigators will give two sessions of iTBS separated by 15 min.
  Arms: active and active
Device: sham and active TBS — The investigators will perform standard intermittent TBS (iTBS) parameters to left DLPFC of every patient in the study. The frequency parameters of TBS are 3-pulse 50- Hz bursts, every 200 ms at 5 Hz, and the intensity is 90% of active motor threshold. A single session of iTBS contains 2 s of TBS repeated every 10 s for 20 times. In this study, The investigators will give two sessions of iTBS separated by 15 min. Sham stimulation applies the same iTBS protocol with the sham coil.
  Arms: sham and active

SUMMARY:
This is a pilot study to identify a homogeneous cohort of pathologically specific dementia with SNAP for clinical trial of brain stimulation.

DETAILED DESCRIPTION:
The investigators apply the NIA-AA criteria to identify the individuals of biomarker-defined SNAP endophenotype. This is a prospective, randomized controlled clinical trial for the first two weeks, followed by an open-label trial for the next two weeks, and combined functional neuroimaging study of 18F-FDG-PET to further explore the potential mechanisms. A total of 20 SNAP dementia patients will be recruited for consecutive two years, and be subjected to iTBS for 5 daily interventions per week for four consecutive weeks. Cognitive evaluation will be performed before and immediately after TBS intervention, and 8 weeks after TBS. Data on functional neuroimaging will be also collected before and after TBS protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 50-90 year.
2. Patients meet NIA-AA research criteria for suspected non-Alzheimer disease pathophysiology (SNAP) (Petersen, Smith et al. 1999; Jack, Bennett et al. 2018), and DSM-5 criteria for major neurocognitive disorder of dementia (Regier, Narrow et al. 2013).
3. Amyloid PET should ever be performed.
4. The CDR of subjects can be 0.5-2.

Exclusion Criteria:

1. Any subject has a definite diagnosis of epilepsy or history of seizure attack.
2. Current or past history of clinically significant neurological insults affecting brain structure or function like completed stroke, head injury or brain tumor. (cerebrovascular disorders, hydrocephalus and intra-cranial mass, documented by MRI; a history of traumatic brain injury or another neurological disease).
3. Any subject has clinically significant or unstable medical diseases including metabolic, renal, liver, lung or cardiovascular disorders including metabolic, renal, liver, lung or cardiovascular disorders.
4. Any subject has current alcohol or other substances abuse and/ or dependence within the recent one year, or prolonged history of major psychiatric disorder like schizophrenia, bipolar disorder, and previously prolonged substances abuse.
5. Any females who is pregnant or lactating.
6. General MRI, TMS and/or PET exclusion criteria including subjects who had received brain aneurysm surgery, or implanted pacemaker, mechanical valves, cochlear implant or other metal devices/ objects that are not MR compatible in the body.

Withdrawal criteria

1. Complications onset after intervention that affect efficacy and safety judgments.
2. New onset or progression of disease that may affect outcomes.
3. Use of other therapies or drugs during the intervention period to change cognitive functions.
4. Any subjects who are recognized as high risk of adverse effects by principle investigator.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The changes of Mini-Mental State Examination (MMSE) total scores | baseline (T0) and immediately after 2 weeks of TBS (T2), and 4 weeks of TBS (T4), and 8-week follow-up after TBS (T12)
  The changes of Mini-Mental State Examination (MMSE) total scores (score range from 0 to 30, higher values represent a better cognitive outcome)
The changes of Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog) total scores | baseline (T0) and immediately after 2 weeks of TBS (T2), and 4 weeks of TBS (T4), and 8-week follow-up after TBS (T12)
  The changes of Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog) total scores (score range from 0 to 70, higher score indicates a worse cognitive outcome)

SECONDARY OUTCOMES:
The standard uptake values changes of FDG-PET | baseline (T0) and immediately after 2 weeks of TBS (T2), and 4 weeks of TBS (T4)
  The standard uptake values (SUV) changes of cerebral glucose metabolism using 18F-FDG-PET

CONTACTS AND LOCATIONS:
Overall Officials: KUAN YI WU, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Guishan, Taiwan